CLINICAL TRIAL: NCT05934747
Title: Aim 3 Particle Swarm Optimization Postural Instability Gait Disorder
Brief Title: Aim 3 Particle Swarm Optimization PIGD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00019089
Record Dates: First submitted 2023-06-28; First posted 2023-07-07 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Parkinson's Disease and Parkinsonism
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: DBS — Deep Brain Stimulation

SUMMARY:
In Parkinson's disease (PD) patients undergoing standard-of-care Deep Brain Stimulation (DBS) therapy, to compare the effect on Parkinson's symptoms of two different neurostimulator settings designed to differ from each other as much as possible with respect to how much they activate two different neuroanatomical structures: the axonal pathway from Globus Pallidus (GP) to Pedunculopontine Nucleus (PPN), and the axonal pathway from PPN to GP.

DETAILED DESCRIPTION:
In Parkinson's disease (PD) patients undergoing standard-of-care Deep Brain Stimulation (DBS) therapy, to compare the effect on Parkinson's symptoms of two different neurostimulator settings designed to differ from each other as much as possible with respect to how much they activate two different neuroanatomical structures: the axonal pathway from Globus Pallidus (GP) to Pedunculopontine Nucleus (PPN), and the axonal pathway from PPN to GP. In this respect, the present protocol is similar to Protocol STUDY00008644. In fact, that protocol, and this one, cover different Aims of the same NIH-funded project. Protocol STUDY00008644 tested different neurostimulor settings for a few hours in the laboratory only; the present protocol also tests them for two weeks between laboratory testing sessions. This is essential, for several reasons. First, clinically relevant outcome measures, such as ADL (activities of dailly life) and QOL (quality of life) scales require observation for longer than a few hours in the laboratory. Second, DBS effects are not instantaneous, and prolonged observation is required to determine the full effect of neurostimulator settings. Third, we intend, if our hypothesis is confirmed (that activation of the PPN-to-GP pathway is most effective for the postural-instability / gait-disorder (PIGD) complex) to propose a clinical trial of neurostimulator settings designed to maximize activation of this pathway; the present protocol will yield data and experience essential for designing and proposing such a trial.

ELIGIBILITY:
* Diagnosis of Parkinson's Disease
* Bilateral DBS in STN or GP
* At least 3 months after lead implantation
* Montreal Cognitive Assessment (MoCA):

MoCA=23+

OR: If MoCA score is 23 or less, UBACC will be performed to ensure capacity to consent. If UBACC results are unclear, the MacCAT-CR will be performed. Failed or unclear MacCAT-CR results will exclude the study candidate.

* Between 18-85 years of age
* Has undergone pre-operative 7T MRI (as part of protocol #1210M22183 or standard-of-care) and post-operative CT imaging (standard of care).

8.2 Exclusion Criteria:

* Inability to walk in the off-med, off-stimulation condition (even with safety harness)
* Gait impaired significantly by a condition other than PD
* Breaks or shorts in active contacts
* IPG battery nearing end of life (in patients with primary-cell IPGs)
* Females who are nursing or pregnant

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-19 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Unified Parkinson's Disease Rating Scale Movement Disorders Society revision, MDS-UPDRS | 1 hour and 2 weeks after intiating stimulation
  Difference in scores on MDS-UPDRS

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States